CLINICAL TRIAL: NCT02108860
Title: Abatacept (CTLA4-Ig) for the Treatment of Relapsing, Non-Severe, Granulomatosis With Polyangiitis (Wegener's) (ABROGATE)
Brief Title: Abatacept for the Treatment of Relapsing, Non-Severe, Granulomatosis With Polyangiitis (Wegener's)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: The Cleveland Clinic (Other); Bristol-Myers Squibb (Industry); University of Pennsylvania (Other); National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABROGATE 5527; 2013-005535-24 (EudraCT Number); U54AR057319 (NIH)
Record Dates: First submitted 2014-03-27; First posted 2014-04-09 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Granulomatosis With Polyangiitis (Wegener's); Granulomatosis With Polyangiitis; Wegener's Granulomatosis; ANCA-Associated Vasculitis
Keywords: Granulomatosis with polyangiitis (Wegener's); Granulomatosis with polyangiitis; GPA; Wegener's granulomatosis; Wegener granulomatosis; Anti Neutrophil Cytoplasmic Antibody Associated Vasculitis; ANCA Associated Vasculitis; AAV; Vasculitis; Systemic vasculitis; Systemic inflammatory disease; Lung Diseases; Respiratory Tract Diseases; Vascular Diseases; Abatacept; CTLA4-Ig; Immunosuppressive agent; Prednisone; Glucocorticoids; Glucocorticoid; Corticosteroid; Corticosteroids; Treatment; Pharmacologic Actions; Therapeutic Uses; Anti Inflammatory Agents
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis; Systemic Vasculitis; Lung Diseases; Respiratory Tract Diseases; Vascular Diseases | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Blinded abatacept (Experimental): Participants will receive blinded abatacept 125 mg administered by subcutaneous injection once a week for at least 12 months. Subjects may be removed from treatment earlier due to a disease relapse, disease worsening, or if they have not achieved remission by treatment month 6.
  Interventions: Drug: Abatacept
- blinded placebo (Placebo Comparator): Participants will receive blinded placebo. Placebo will be administered by subcutaneous injection once a week for at least 12 months. Subjects may be removed from treatment earlier due to a disease relapse, disease worsening, or if they have not achieved remission by treatment month 6.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Abatacept — Those randomized to abatacept will receive abatacept 125 mg administered by subcutaneous injection once a week Participants randomized to either the abatacept or the placebo arm who experience a non-severe disease relapse, non-severe disease worsening, or who have not achieved remission by month 6 will have the option of entering an open-label trial period whereby they would receive open-label abatacept. .
  Other Names: CTLA4-Ig; Orencia
  Arms: Blinded abatacept
Drug: placebo — Those randomized to placebo will receive a sterile placebo solution administered by subcutaneous injection once a week.
  Arms: blinded placebo

SUMMARY:
Multi-center, randomized, double-blind, placebo-controlled trial to evaluate the efficacy of abatacept to achieve sustained glucocorticoid-free remission in patients with relapsing non-severe granulomatosis with polyangiitis (Wegener's) (GPA) . Participants will be randomized 1:1 to receive either abatacept 125 mg or placebo administered by subcutaneous injection once a week. Participants will continue on study treatment for a minimum of 12 months unless they experience a disease relapse or disease flare.

Participants who experience a non-severe disease relapse, non-severe disease worsening, or who have not achieved remission by month 6 will have the option of entering an open-label trial period whereby they would receive open-label abatacept.

DETAILED DESCRIPTION:
Multi-center, randomized, double-blind, placebo-controlled trial to evaluate the efficacy of abatacept to achieve sustained glucocorticoid-free remission in patients with relapsing non-severe GPA. Patients who enter the trial will be maintained on a stable dose of their maintenance immunosuppressive agent which may include methotrexate (MTX), azathioprine (AZA), or mycophenolate (MA) and will undergo a blinded randomization to receive abatacept or placebo. Patients will additionally receive prednisone 30 mg daily that will then be tapered to zero using a standardized tapering schedule.

If an enrolled patient experiences a non-severe relapse or non-severe disease worsening though common closing, or if they have not achieved remission by month 6, they will have the option of entering an open-label trial period whereby they would receive abatacept in conjunction with their maintenance immunosuppressive and a standardized glucocorticoid taper. Patients with a severe disease relapse or severe disease worsening will have met criteria for early termination criteria and be removed from active study treatment. Patients will remain on study until reaching criteria for early termination or until common closing, 12 months after randomization of the final patient. After common closing or early termination, patients will be treated with best medical judgment and will undergo a post-treatment safety visit 3 months after coming off of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be considered as being best characterized as GPA and not microscopic polyangiitis (MPA) or eosinophilic granulomatosis with polyangiitis (EGPA) and must have met at least 2 of the 5 modified ACR classification criteria for GPA. These do not need to be present at the time of study entry. The modified ACR criteria are:

   1. Nasal or oral inflammation, defined as the development of painful or painless oral ulcers or purulent or bloody nasal discharge
   2. Abnormal chest radiograph, defined as the presence of nodules, fixed infiltrates, or cavities
   3. Active urinary sediment, defined as microscopic hematuria (>5 red blood cells per high power field) or red blood cell casts
   4. Granulomatous inflammation on biopsy, defined as histologic changes showing granulomatous inflammation within the wall of an artery or in the perivascular or extravascular area (artery or arteriole)
   5. Positive anti-neutrophil cytoplasmic antibody (ANCA) test specific for proteinase-3 or myeloperoxidase measured by enzyme-linked immunoassay
2. Relapse of GPA within the 28 days prior to screening where the active disease features meet the following definition of non-severe disease:

   1. No disease manifestations that would be scored as a major element in the BVAS/WG
   2. Absence of any disease feature that poses an immediate threat to either a critical individual organ or the patient's life
3. Age 15 and older
4. Willing and able to comply with treatment and follow-up procedures
5. Both women and men must be willing to use an effective means of birth control while receiving treatment through this study. Women should continue the use of an effective means of birth control for a minimum of 14 weeks after the last dose of study drug. Effective contraception methods include abstinence, oral contraceptives (birth control pills), IUD, diaphragm, Norplant, approved hormone injections, condoms, or medical sterilization. If applicable, participating sites will defer to their local authorities if they require stricter guidelines on the types of allowable contraception methods.
6. Willing and able to provide written informed consent (and written assent of minor participants if applicable.)

Exclusion Criteria:

1. Presence of involvement that does not meet the criteria for non-severe disease
2. Treatment with CYC within 3 months prior to screening
3. Treatment with methylprednisolone 1000 mg within 28 days prior to enrollment
4. Treatment with prednisone or prednisolone> 30 mg/day for > 28 days immediately prior to study entry
5. Initiation or dose increase of the maintenance immunosuppressive agent (MTX, AZA, MA) within 3 months prior to screening
6. Evidence of active infection (includes chronic infection)
7. Patients who are pregnant or who are nursing
8. Known infection with human immunodeficiency virus (HIV), hepatitis C, or a positive hepatitis B surface antigen
9. Inability to comply with study guidelines
10. Cytopenia: platelet count < 100,000/mm3, white blood cell count (WBC) < 3,000/mm3 (3 x 109/L), absolute neutrophil count < 1500/mm3, hemoglobin (Hgb) < 8.5 g/dL
11. Chronic renal insufficiency defined by a creatinine clearance of less than or equal to 20 ml/min
12. AST or ALT > 3 times above the upper limit of the normal laboratory range
13. Known current use of illegal drugs
14. Other uncontrolled disease (co-morbidity) that could prevent a patient from fulfilling the study requirements or that would substantially increase the risk of study procedures
15. History of malignancy within the past five years or any evidence of persistent malignancy, except fully excised basal cell or squamous cell carcinomas of the skin, or cervical carcinoma in situ which has been treated or excised in a curative procedure
16. Receipt of an investigational agent or device within 30 days prior to enrollment or 5 half lives of the investigational drug (whichever is longer)
17. A live vaccination fewer than 3 months before enrollment
18. Current clinical, radiographic, or laboratory evidence of active tuberculosis
19. A history of active tuberculosis within the past 3 years even if treated
20. A history of active tuberculosis greater than 3 years ago unless there is documentation of prior anti-tuberculosis treatment of appropriate duration and type
21. Latent tuberculosis unless there is documentation of prior anti-tuberculosis treatment of appropriate duration and type
22. Latent tuberculosis currently being treated with isoniazid (INH) or other therapy for latent tuberculosis given according to local health authority guidelines (e.g., Center for Disease Control (CDC)) who have received such therapy for 4 weeks or less prior to randomization (Day 1). Subjects with a positive tuberculosis screening test indicative of latent tuberculosis will be eligible for the study if they have no evidence of current tuberculosis on chest xray at screening and they are actively being treated for tuberculosis with INH or other therapy for latent tuberculosis given according to local health authority guidelines (e.g., CDC) that has been given for at least 4 weeks prior to randomization (Day 1). These subjects must complete treatment according to local health authority guidelines.
23. History of herpes zoster that resolved less than 2 months prior to enrollment
24. Treatment with rituximab or any other biologic B cell depleting agent within the past 6 months
25. Treatment with alemtuzumab or anti-thymocyte globulin within the last 12 months
26. Treatment with intravenous immunoglobulin given at an immunomodulatory dosage or plasma exchange within the past 3 months. Patients can be enrolled if they are otherwise eligible and receiving immunoglobulin replacement for hypogammaglobulinemia.
27. Treatment with infliximab, etanercept, adalimumab, tocilizumab, or any other biologic agent within the past 3 months or 5 half lives of the agent (whichever is longer)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-04-25 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Ability of abatacept to reduce the treatment failure rate | 12 months
  Treatment failure will be defined as relapse, disease worsening, or failure to achieve a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) = 0 or 1 by 6 months.
  Relapse will be defined as any of the following after remission: an increase in BVAS/WG, development of a new BVAS/WG item, or symptoms/signs of GPA that cannot be attributed to any cause other than GPA and that requires institution or dosage increase of prednisone.
  Disease worsening will be defined as any of the following prior to remission: an increase in BVAS/WG, development of a new BVAS/WG item, or symptoms/signs of GPA that cannot be attributed to any cause other than GPA and that requires institution or dosage increase of prednisone.

SECONDARY OUTCOMES:
Duration of glucocorticoid-free periods | 12 months
  Effect of abatacept on increasing duration of glucocorticoid-free periods for participants. Patients will be treated with abatacept for a minimum of 12 months unless they reach study criteria for early termination or until common closing. Common closing will be 12 months after randomization of the final patient.
Severity of relapses in those treated with abatacept versus placebo | 12 months
  Severity of GPA disease relapses in those treated with abatacept versus placebo. Patients will be treated with abatacept for a minimum of 12 months unless they reach study criteria for early termination or until common closing. Common closing will be 12 months after randomization of the final patient.
Health-related quality of life in those treated with abatacept versus placebo | 12 months
  Health-related quality of life in those treated with abatacept versus placebo as assessed using the SF-36 and PROMIS questionnaires. Patients will be treated with abatacept for a minimum of 12 months unless they reach study criteria for early termination or until common closing. Common closing will be 12 months after randomization of the final patient.
Prevention of disease- or treatment-related damage with abatacept versus placebo | 12 months
  Prevention of disease or treatment related damage as assessed by the infection rate in both treatment arms. Patients will be treated with abatacept for a minimum of 12 months unless they reach study criteria for early termination or until common closing. Common closing will be 12 months after randomization of the final patient.
Safety of abatacept in GPA | 12 months
  Safety of abatacept in patients with GPA as assessed by reported adverse events. Patients will be treated with abatacept for a minimum of 12 months unless they reach study criteria for early termination or until common closing. Common closing will be 12 months after randomization of the final patient.

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Langford, MD, MHS, Principal Investigator — The Cleveland Clinic; Jeffrey P Krischer, PhD, Principal Investigator — University of South Florida; Peter A Merkel, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (20):
- United States (10):
  - Cedars Sinai Medical Center, Los Angeles, Los Angeles, California
  - University of South Florida Rheumatology, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, St. Paul's Rheumatology Clinic, Vancouver, British Columbia
  - St. Joseph's Hospital, Hamilton, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Toronto, Ontario
- Medius Kliniken, Kirchheim unter Teck, Germany
- St. Vincent's University Hospital, Dublin, Ireland
- United Kingdom (4):
  - University of Aberdeen, Aberdeen
  - University of Cambridge- Addenbrookes Hospital, Cambridge
  - Nottingham University Hospitals, Nottingham
  - Royal Berkshire Hospital, Reading

REFERENCES:
- [Derived] Hung W, Cusnir I, Habib S, Smylie M, Solez K, Yacyshyn E. Immune checkpoint inhibitor-induced granulomatosis with polyangiitis. Rheumatology (Oxford). 2021 Jun 18;60(6):e190-e191. doi: 10.1093/rheumatology/keaa818. No abstract available. PMID 33367837